CLINICAL TRIAL: NCT05790863
Title: Effects of Low-volume High-intensity Training Versus Moderate-intensity Continuous Training on Physical Performance in Older Adults With Possible Sarcopenia
Brief Title: Effects of Low-volume HIIT Versus MICT on Physical Performance in Older Adults With Possible Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20221231001
Record Dates: First submitted 2023-03-02; First posted 2023-03-30 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity interval training group (Experimental): Each ergometer cycling training session consists of a warm-up phase lasting two minutes, five interval bouts of one minute each at 77% to 90% of one's HRmax, separated by one minute of passive or low-intensity recovery, and a three-minute cool-down phase. After 4 weeks of the intervention, the minimal intensity that had to be met will be progressively raised (weeks 1-4: 76-85%, weeks 5-7: 85-90%HRmax, respectively). For individuals who are unable to reach 77% HRmax, scores of 15 to 17 (hard to very hard) on the Borg scale will be followed.
  Interventions: Device: Ergometer cycling
- Moderate-intensity continuous training group (Active Comparator): During the first four weeks, participants will be advised to modify the pedal cadence and/or resistance of the ergometer to obtain an HR equivalent to 65-70% HRmax, rising to 70-76% HRmax during the final 3 weeks. Each session lasts less than 25 minutes of moderate-intensity continuous ergometer cycling, which starts with a two-minute warm-up and ends up with a three-minute cool-down.
  Interventions: Device: Ergometer cycling

INTERVENTIONS:
Device: Ergometer cycling — Paticipants will receive 21 sessions (3 sessions/week) of training for 7 weeks with the arm-leg cycle ergometer (SCIFIT, REX7000, US)

SUMMARY:
Background: Sarcopenia is an age-related geriatric syndrome characterized by progressive loss of muscle mass and function. Before the diagnosis of sarcopenia, a "possible sarcopenia" stage has been proposed recently, characterized by low muscle strength or poor physical performance, even with normal muscle mass. The definition of "possible sarcopenia" emphasizes the importance of early intervention. Due to the lack of effective pharmaceutical treatments, exercise is recommended as the most available intervention for sarcopenia. High-intensity interval training (HIIT), a time-efficient aerobic training, has gained increasing popularity for its benefits in physiologic outcomes such as muscle strength and physical functions in other populations. However, the benefits of HIIT have not been well-studied following older adults with possible sarcopenia. In the present study, we aim to investigate the effects of a 7-week HIIT and moderate-intensity continuous aerobic training (MICT) on physical performance in older individuals with possible sarcopenia. We hypothesize that HIIT will confer physical benefits over MICT (i.e., traditional endurance exercise) and will be generally well-tolerated in older adults.

Method: The participants will be randomly allocated into the HIIT or MICT group (1:1 ratio). The participants will receive the training 3 times per week over seven weeks. HIIT consists of 5 bouts of interval training intensity with 1-minute-high intensity (76-90% HRmax) and 1-minute recovery per session (total 15 minutes with warm-up and cool-down). MICT will adopt an intensity of 65-70% HRmax training that lasts less than 30 minutes per session (total 25 minutes with warm-up and cool-down). Evaluation will be performed at baseline, after 4 weeks, and 7 weeks of the intervention. The primary outcomes include 10-meter walking test and the five-time chair stand test. The secondary outcomes include grip strength, the functional stretch test; the Exercise Enjoyment Scale and the Physical Activity Enjoyment Scale for affective valence.

Discussion: This is the first study to investigate the effects of low-volume HIIT on physical performance and affective valence in older adults with possible sarcopenia. This study will provide critical evidence to guide early prevention and intervention of exercise regimens for possible sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 60 years or older, living in the community
* Able to walk with or without assistive devices
* Recovery from COVID-19 over two months
* With a preliminary screening of SARC-F score ≥4 or calf circumference less than 34cm for man, 33cm for woman will be invited to strength and physical performance measurement
* Handgrip strength less than 28 kg for man, 18 kg for woman and/or gait speed<1m/s and/or 5-time chair stand test ≥12 s.

Exclusion Criteria:

* Inability to undertake exercise due to neuromuscular and/or musculoskeletal limitations
* Uncontrolled hypertension (systolic BP>170 or diastolic BP>100 mmHg)
* Reported chronic cardiopulmonary insufficiency in medical history
* Reported vital organ failure and malignancy in medical history
* Cognitive impairments (mini-mental test score<21) with low compliance
* History of lower limb surgeries, fractures, neurological problems, systemic problems, and any other contraindications for aerobic training will be excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in time of the The 5 repeated sit-to-stand test after 7 weeks of intervention | Baseline and after 7 weeks of intervention
  The 5 repeated sit-to-stand test is a validated way to reflect the lower limb muscle strength and balance ability of the elderly. Subjects are required to complete 5 times of standing up and sitting down as fast as possible without using handrails or other assistance by crossing the arms in front of the chest. Care should be taken to ensure that the knee joints are completely straight before sitting down. The time of completing test will be recorded.
  Change=(week 7 time- baseline time)

SECONDARY OUTCOMES:
Change from Baseline in walking speed of the 10 meter-walk test after 7 weeks of intervention | Baseline and after 7 weeks of intervention
  A 10-meter track needs to be marked before measurement, with separate markers at 2 meters and 8 meters. Timing starts when the subject's front foot crosses the 2-meter marker and ends at 8 meters. Subjects will be allowed to use walking aids, but no assistance will be allowed. Three tests will be performed with a 1-minute break in between; the average walking speed will be calculated.
  Change=(week 7 speed- baseline speed)
Change from Baseline in Hand grip strength after 7 weeks of intervention | Baseline and after 7 weeks of intervention
  Subjects will be instructed to take a seat measurement with their arm extended, forearm unsupported, elbow flexed at 90 degrees, wrist in a neutral position, and grip tightened to maximum capacity by using a Jamar dynamometer. The dominant hand will perform the grip strength twice, and the maximum force will be recorded.
  Change=(week 7 strength- baseline stength)
Change from Baseline in distance of The functional stretch test after 7 weeks of intervention | Baseline and after 7 weeks of intervention
  The subject stands sideways against the wall with the arm elevated and parallel, reaches forward as far as possible with the body balanced, keeping the feet unmoving. The distance of forward extension reach of the middle finger end position will be measured twice, with a rest interval of 1 minute, and the average value will be obtained.
  Change=(week 7 score- baseline score)
Change from Baseline in score of The Exercise Enjoyment Scale after 7 weeks of intervention | Baseline and after 7 weeks of intervention
  EES is a single-item 7-point scale with the following instruction: "Please measure how much you are enjoying the current exercise." It ranges from "1" (not at all enjoyable) to "7" (extremely enjoyable) Change=(week 7 score- baseline score)
Change from Baseline in score of The Physical activity enjoyment scale after 7 weeks of intervention | Baseline and after 7 weeks of intervention
  PACES has 18 different items on a 7-point scale, is used to quantify post-exercise satisfaction (e.g., "1" I enjoyed the sport, "7" I hated the sport). "Please rate how you feel about the activity you just completed" is the directive.
  Change=(week 7 score- baseline score)

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Brain Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Reljic D, Frenk F, Herrmann HJ, Neurath MF, Zopf Y. Effects of very low volume high intensity versus moderate intensity interval training in obese metabolic syndrome patients: a randomized controlled study. Sci Rep. 2021 Feb 2;11(1):2836. doi: 10.1038/s41598-021-82372-4. PMID 33531522
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Rosenberg IH. Sarcopenia: origins and clinical relevance. J Nutr. 1997 May;127(5 Suppl):990S-991S. doi: 10.1093/jn/127.5.990S. PMID 9164280
- [Background] Dent E, Morley JE, Cruz-Jentoft AJ, Arai H, Kritchevsky SB, Guralnik J, Bauer JM, Pahor M, Clark BC, Cesari M, Ruiz J, Sieber CC, Aubertin-Leheudre M, Waters DL, Visvanathan R, Landi F, Villareal DT, Fielding R, Won CW, Theou O, Martin FC, Dong B, Woo J, Flicker L, Ferrucci L, Merchant RA, Cao L, Cederholm T, Ribeiro SML, Rodriguez-Manas L, Anker SD, Lundy J, Gutierrez Robledo LM, Bautmans I, Aprahamian I, Schols JMGA, Izquierdo M, Vellas B. International Clinical Practice Guidelines for Sarcopenia (ICFSR): Screening, Diagnosis and Management. J Nutr Health Aging. 2018;22(10):1148-1161. doi: 10.1007/s12603-018-1139-9. PMID 30498820
- [Background] Lozano-Montoya I, Correa-Perez A, Abraha I, Soiza RL, Cherubini A, O'Mahony D, Cruz-Jentoft AJ. Nonpharmacological interventions to treat physical frailty and sarcopenia in older patients: a systematic overview - the SENATOR Project ONTOP Series. Clin Interv Aging. 2017 Apr 24;12:721-740. doi: 10.2147/CIA.S132496. eCollection 2017. PMID 28490866
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle. Part II: anaerobic energy, neuromuscular load and practical applications. Sports Med. 2013 Oct;43(10):927-54. doi: 10.1007/s40279-013-0066-5. PMID 23832851
- [Background] Hannan AL, Hing W, Simas V, Climstein M, Coombes JS, Jayasinghe R, Byrnes J, Furness J. High-intensity interval training versus moderate-intensity continuous training within cardiac rehabilitation: a systematic review and meta-analysis. Open Access J Sports Med. 2018 Jan 26;9:1-17. doi: 10.2147/OAJSM.S150596. eCollection 2018. PMID 29416382
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Mehmet H, Yang AWH, Robinson SR. What is the optimal chair stand test protocol for older adults? A systematic review. Disabil Rehabil. 2020 Oct;42(20):2828-2835. doi: 10.1080/09638288.2019.1575922. Epub 2019 Mar 24. PMID 30907166